CLINICAL TRIAL: NCT04491773
Title: Evaluation of Retinal and Choriocapillary Vascular Changes Using Optical Coherence Tomography Angiography in Patients Undergoing Tadalafil 20mg on Alternative Days for More Than 6 Months: a Single-centre Prospective-control
Brief Title: Study of Retinal and Choriocapillary Vascular Changes in Patients Undergoing Tadalafil 20mg for More Than 6 Months
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1516/19
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2019-11

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing Tadalafil: Patients after radical prostatectomy, undergoing Tadalafil 20 mg orally, on alternative days, for more than 6 months
  Interventions: Drug: Tadalafil 20 MG
- Control Group: Healthy controls without previous surgery of radical prostatectomy.

INTERVENTIONS:
Drug: Tadalafil 20 MG — To study retinal and choriocapillary features in patients undergoing Tadalafil 20 mg orally, on alternate days, for more than 6 months.
  Other Names: Cialis
  Groups: Patients undergoing Tadalafil

SUMMARY:
This study evaluates the retinal and choriocapillary vascular features in patients under the effects of Tadalafil 20mg for more than 6 months, using optical coherence tomography angiography.

DETAILED DESCRIPTION:
Tadalafil is a an inhibitor of the enzyme phosphodiesterase and it works by increasing blood flow to the penis thus promoting the erection.

This drug represents an treatment for erectile dysfunction in patients after radical prostatectomy.

The optical coherence tomography angiography represents a novel and noninvasive diagnostic technique that allows a detailed and quantitative analysis of retinal and choriocapillary vascular features.

The study evaluates the changes in optical coherence tomography angiography features after the somministration of Tadalafil 20 mg orally for more than 6 months.

ELIGIBILITY:
Inclusion Criteria:

* age older than 45 years
* diagnosis of erectile dysfunction due to surgery of radical prostatectomy
* treatment-naïve with Tadalafil for erectile dysfunction for more than 6 months
* absence of diabetes, heart diseases, hypertension
* absence of drug intake
* absence of vitreoretinal, vascular retinal diseases
* absence of previous ocular surgery and congenital eye diseases.
* absence of errors of refraction
* absence of lens opacities
* absence of low-quality OCT and OCTA images

Exclusion Criteria:

* age younger than 45 years
* diagnosis of erectile dysfunction due to other causes
* previous treatments before Tadalafil for erectile dysfunction
* presence of diabetes, heart diseases, hypertension
* drug intake
* vitreoretinal and vascular retinal diseases
* previous ocular surgery and congenital eye diseases
* errors of refraction
* lens opacities
* low-quality OCT and OCTA images

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participans were older than 45 years with diagnosis of erectile dysfunction due to surgery of radical prostatectomy. They did not receive previous treatment before Tadalafil. They did not present any ophthalmological disease, diabetes, heart diseases and hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal and choriocapillary vessel density in patients undergoing Tadalafil for more than 6 months | More than 6 months
  Changes in retinal and choriocapillary vessel density in patients after radical prostatectomy, undergoing Tadalafil 20 mg orally on alternate days for more than 6 months, using optical coherence tomography angiography.
  The parameters analyzed by optical coherence tomography angiography were: retinal and choriocapillary vessel density

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy